CLINICAL TRIAL: NCT06727149
Title: The Effect of Using Virtual Reality on Pain, Fear and Anxiety by School-Age Children During Venipuncture: A Randomized Controlled Study
Brief Title: The Effect of Virtual Reality on Pain, Fear and Anxiety by Children During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02082022
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pain; Fear; Anxiety
Keywords: pain management; pain in children; fear in children; anxiety; virtual reality
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Procedure) (Experimental)
  Interventions: Other: Control Group
- Virtual Reality Group (Experimental)
  Interventions: Other: Virtual Reality Group

INTERVENTIONS:
Other: Control Group — No intervention was performed to reduce pain, fear and anxiety in the control group
  Arms: Control Group (Standard Procedure)
Other: Virtual Reality Group — The children in the VR group were informed about the virtual reality glasses and told that they could remove the glasses at any time if they felt uncomfortable during the procedure
  Other Names: Experimental
  Arms: Virtual Reality Group

SUMMARY:
There are many approaches to reduce pain, fear and anxiety that may occur in children during invasive procedures. The most commonly used of these approaches is virtual reality, which is a method of distracting attention and designed with cognitive and behavioral techniques. This study was conducted in a randomized controlled experimental design to determine the effect of virtual reality glasses given to children during venepuncture on pain, fear and anxiety.

The research was conducted between September 2022 and May 2023 with two parallel groups in the pediatric inpatient service of a private hospital in western Turkey. The study sample consisted of children aged 6-12 years and the sample was randomization, the control group (n=30) and the virtual training group (30) constituted a total of 60. The data of the study were obtained from Child Information Form, Wong-Baker Faces Pain Rating Scale, State-Trait Anxiety Inventory for children. The data were analyzed using SPSS 25 program.

DETAILED DESCRIPTION:
This randomized controlled clinical trial (RCT) was conducted between September 2022 and May 2023 with two parallel groups in the pediatric inpatient service of a private hospital in western Turkey.

In order to determine the number of patients constituting the research sample, a similar study in the relevant literature was taken as an example and the power analysis G*Power 3.1 software was used. In this study, in order to reach a power level of 95% at a 0.5 effect size and 5% error level, the sample size was calculated as 56, with 28 participants in each group. Considering the high power of the test and the losses in the study, a total of 60 people were reached, 30 in each group.The study sample consisted of children aged 6-12 years with stable hemodynamics who were undergoing venipuncture, had sufficient cognitive and communication abilities to rate their pain, fear, and anxiety levels, and were willing to participate. This group was selected because children of that age are the most cooperative. All participating children gave verbal consent to participate, and their families provided written consent. Children with unstable conditions and vital signs, intubated, had visual problems or did not want to participate in the study were excluded.

Children meeting the sampling criteria were randomly allocated to one of the two groups: the VR group and the control group. First, group numbers were written on uniform pieces of paper as 30 VR 30 control, and the papers were placed into closed box. Participants were asked to pick one card among the 60. They were assigned to the group according to their card. Thus, each group had 30 children in each group and 60 children in the study.

The research's outcomes were pain levels assessed with the Wong-Baker Faces Pain Rating Scale (WBS), fear levels assessed with the Children's Fear Scale (CFS), anxiety levels assessed with the State-Trait Anxiety Inventory for children (STAI-CH). WBS and CFS were scored separately by the researcher, the child and the parent, and STAI-CH was scored by the child alone within five minutes before and immediately after the procedure. All ratings were done blindly to ensure that the observers did not influence each other's scores.

The researchers created the child information form and included nine questions about the children's age, sex, parents' age, education level, economic level, and type of family.

Procedure One researcher (İ.A.) provided information about the study to the children and their parents in the patient rooms. Children who met the inclusion criteria were included in the study and informed consent forms were obtained from the child and parent. Participants were randomly assigned to the groups. The child information form was filled out. The WBS and CFS were obtained from the child and parent by another researcher (G.A.), and the STAI-CH was obtained from the child. Researcher İ.A. scored the WBS and CFS blindly to the child and parent's responses. The children were told that intravenous access would be established and that they would be asked to assess their fear and anxiety with the CFS and STAI-CH immediately before the procedure. The instructions regarding the scales were read to the children. The children scored on paper. Then, the child's parent was asked to score the CFS according to the child's fear. The child and parent did not see each other's scores. Researcher İ.A. scored the CFS. Researcher G.A. was not blinded to the children's and parents' scores.

All children were allowed to have their families with them during the vascular access procedure. The vascular access procedure was performed by the same person in all groups (H.K.). The researcher introduced the materials to the child. After the child gave permission by asking, "Which arm can I open the vascular access in?", the researcher performed the vascular access procedure. If the procedure was unsuccessful, the child was asked for permission to use the other arm. If the child did not want the vascular access immediately, a period of time was waited. When the child was ready, the researcher performed the procedure again. The children in the VR group were informed about the virtual reality glasses and told that they could remove the glasses at any time if they felt uncomfortable during the procedure (Researcher İ.A.). Before the vascular access procedure began, the children were given VR glasses (Oculus Quest 2) and were allowed to watch the three-dimensional video until the procedure was completed. No intervention other than the standard procedure was performed on the children in the control group during the vascular access procedure. In both groups, the child, parent, and researcher (İ.A.) scored the WBS and CFS blindly to each other immediately after the procedure. The child was also asked to score the STAI-CH.

Data analysis The data obtained in the study were analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Descriptive statistical methods were used in the evaluation of the data as number, percentage, mean, standard deviation. Differences between the rates of categorical variables in independent groups were analyzed with Chi-Square and Fisher exact tests. T-test was used to compare quantitative continuous data between two independent groups. Dependent groups t-test was used to compare within-group measurements. Relationships between the dependent variables of the study were tested with Pearson correlation and regression analysis. In this study, the reliability of the Wong-Baker Facial Expressions Rating Scale was found to be high as Cronbach's Alpha=0.872, the reliability of the Child Fear Scale as Cronbach's Alpha=0.869, and the reliability of the State Anxiety Scale for Children as Cronbach's Alpha=0.885. Pain; Fear was assessed by the child, parent and researcher and the agreement between the assessments was found to be high (Kappa (κ) =0.789, p=0.000). Fear was assessed by the child, parent and researcher and the agreement between the assessments was found to be high (Kappa (κ) =0.816, p=0.000).

ELIGIBILITY:
Inclusion Criteria:

The children

* who were aged between 6-12 years
* were healty
* stable hemodynamics who were undergoing venipuncture
* who were sufficient cognitive and communication abilities to rate their pain, fear, and anxiety levels,
* were willing to participate. All participating children gave verbal consent to participate, and their families provided written consent

Exclusion Criteria:

* Children with unstable conditions and vital signs, intubated, had visual problems or did not want to participate in the study were excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
pain severity | 8 month
  The children and parents informed about Wong BakerFaces Pain

SECONDARY OUTCOMES:
Fear levels | 8 month
  The children and parents informed about Children Fears Scale
Anxiety levels | 8 month
  The children and parents informed about STAI

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, Phd RN, Principal Investigator — Istanbul Beykent University
Locations (1):
- Istanbul Beykent University, Istanbul, Turkey (Türkiye)